CLINICAL TRIAL: NCT00826332
Title: Transvaginal or Transabdominal Ultrasound Guided Embryo Transfer- Which is Better?
Brief Title: Transvaginal vs Transabdominal Ultrasound Guided Embryo Transfer
Acronym: TVUSET
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Ariel Revel, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0594-08-HMO-CTIL
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: In Vitro Fertilization
Keywords: ultrasound; IVF; Embryo transfer; Pregnancy rate; female patient undergoing IVF

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abdominal (Active Comparator): Transabdominal ultrasound guided embryo transfer
  Interventions: Procedure: transabdominal ultrasound
- Vaginal (Active Comparator): Transvaginal ultrasound guided embryo transfer
  Interventions: Procedure: transvaginal ultrasound

INTERVENTIONS:
Procedure: transabdominal ultrasound — transabdominal ultrasound
  Arms: Abdominal
Procedure: transvaginal ultrasound — transvaginal ultrasound
  Arms: Vaginal

SUMMARY:
Embryo transfer is the last step in the IVF process. it is now recognized that this step should be done carefully and that it affects success rates. in recent years, sonographic guidance appears to increase success rates.

DETAILED DESCRIPTION:
Embryo transfer is the last step in the IVF process. it involves the insertion of a soft catheter through the uterine cervix. It is now recognized that this step should be done carefully and that it affects success rates. The embyos should be carefully deposited in the cavity. special care should be given to avoid touching the uterine fundus during the procedure. In recent years, sonographic guidance appears to increase success rates.

ELIGIBILITY:
Inclusion Criteria:

* high quality embryos fro transfer

Exclusion Criteria:

* repeated IVF failure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
pregnancy | 14 days

SECONDARY OUTCOMES:
patient satisfaction | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel

REFERENCES:
- [Background] Sallam HN, Sadek SS. Ultrasound-guided embryo transfer: a meta-analysis of randomized controlled trials. Fertil Steril. 2003 Oct;80(4):1042-6. doi: 10.1016/s0015-0282(03)01009-4. PMID 14556831
- [Derived] Karavani G, Ben-Meir A, Shufaro Y, Hyman JH, Revel A. Transvaginal ultrasound to guide embryo transfer: a randomized controlled trial. Fertil Steril. 2017 May;107(5):1159-1165. doi: 10.1016/j.fertnstert.2017.01.023. Epub 2017 Mar 24. PMID 28347493